CLINICAL TRIAL: NCT04931212
Title: Fetoscopic Endoluminal Tracheal Occlusion (FETO) With Smart-TO Device in Fetuses With Congenital Diaphragmatic Hernia and Moderate to Severe Pulmonary Hypoplasia: Proof of Concept and Safety Evaluation.
Brief Title: Fetoscopic Endoluminal Tracheal Occlusion (FETO) With Smart-TO
Acronym: Smart-FETO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-A02834-35; 2020-A02834-35 (Other: ID-RCB)
Record Dates: First submitted 2021-02-06; First posted 2021-06-18 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Congenital Diaphragmatic Hernia
Keywords: Congenital diaphragmatic hernia; Fetal endoscopic tracheal occlusion; Smart-TO balloon; Proof of concept; Safety study
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Procedure: FETO with Smart-TO balloon

INTERVENTIONS:
Procedure: FETO with Smart-TO balloon — Fetal endoscopic tracheal occlusion using the Smart-TO balloon Unplug procedure by peripheral course around the MR scanner
  Other Names: Unplug

SUMMARY:
The purpose of this study is to make the proof of concept and to evaluate the safety of fetoscopic endoluminal tracheal occlusion (FETO) using Smart-TO device in fetuses with congenital diaphragmatic hernia and moderate to severe pulmonary hypoplasia

DETAILED DESCRIPTION:
Congenital diaphragmatic hernia (CDH) leads to lung hypoplasia and impaired lung vasculature. Fetal lung growth may be stimulated by fetal endoscopic tracheal occlusion (FETO). In severe CDH, FETO may improve survival. In the moderate cases, the prematurity induced by the plug-unplug strategy limits the benefit from the lung growth induced by tracheal occlusion.

One of the main drawbacks of FETO is the need for in-utero reversal of tracheal occlusion by the balloon, as the current procedure involves re-establishment of patent airways either electively at 34 weeks' gestation or earlier if required, ideally at least 24 h before birth. Unfortunately, removal of the balloon is a difficult, invasive, and risky procedure. Furthermore, it requires a specialist team to be able to reverse the occlusion at all times. As a result, it is recommended that the patient stays close to a FETO center during the whole duration of the occlusion, which may limit the acceptability of FETO.

The Smart-TO balloon allows an easy, remotely controlled, and non-invasive reversal occlusion, so it allows to overcome issues related to the airway reestablishment. The technology solution is based on a magnetic valve that opens under the influence of the peripheral magnetic field around a magnetic resonance (MR) scanner. The opening of the valve induces the deflation of the balloon, which is then washed out by the fluid coming out from the lungs.

The purpose of this study is to make the proof of concept and to evaluate the safety of fetoscopic endoluminal tracheal occlusion (FETO) using Smart-TO device in fetuses with congenital diaphragmatic hernia and moderate to severe pulmonary hypoplasia. Secondary objectives include evaluation of prematurity, preterm premature rupture of membranes, lung growth, and survival at discharge in case of FETO with Smart-TO balloon.

FETO with Smart-TO balloon will be performed between 27 and 31wks + 6 days depending on the severity of pulmonary hypoplasia, according to the same technique that is used with the balloon usually used for FETO procedure. The unplug procedure will be performed between 34 and 34wks + 6 days or earlier if required. The patient will be asked to make a peripheral course around the MR scanner in order to open the magnetic valve and induce the deflation of the balloon. Ultrasound scan will be performed before and after the unplug procedure, in order to check the balloon did not deflate spontaneously at the time of the unplug, and to check the balloon deflates thanks to the magnetic fringe field of the MR scan. Expelling of the Smart-TO balloon outside the airways will be check at birth by a thorax X-ray.

Patients will be monitored during the whole duration of the study so serious unexpected or adverse reactions can be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or more, who are able to consent, and affiliated to social security
* Singleton pregnancy with fetus with isolated left-sided congenital diaphragmatic hernia (no additional malformation nor chromosomal abnormality) and:

Severe pulmonary hypoplasia defined as observed on expected 'lung-to-head ration' (O/E LHR) <25% irrespective of the liver position as measured between 27wks and 29wks + 6 days Or Moderate pulmonary hypoplasia defined as O/E LHR 25-34.9% (liver up or down) or O/E LHR 35-44.9% with liver up as measured between 30wks and 31wks + 6 days

Exclusion Criteria:

* Maternal contraindication to fetoscopic surgery
* Preterm premature rupture of the membranes (PPROM) or condition strongly predisposing to PPROM or premature delivery
* Impossibility of remain close to the FETO center during the fetal occlusion period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2024-01-14 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Deflation of the Smart-TO balloon after exposure to the fringe field of the MRI | Between 34 and 34+6 amenorrhea weeks
  No visualization of the balloon at ultrasound scan
Expelling of the Smart-TO balloon outside the airways | At birth
  Thorax X-ray of the neonate

SECONDARY OUTCOMES:
Serious unexpected or adverse reactions | From date of inclusion until discharge date from hospitalization of newborn, up 15 months
  Adverse reactions monitoring during the whole study duration
Spontaneous deflation of the balloon | Between the FETO (27amenorrhea weeks) and the unplug procedure (34 amenorrhea weeks)
  Ultrasound scan
Prematurity | At birth
  Gestational age at birth
Preterm premature rupture of the membranes (PPROM) | from date of inclusion until delivery, up to 37 amenorrhea weeks
  Event of PPROM and gestational age at PPROM
Fetal lung growth | Before the unplug procedure
  O/E LHR measurement
Survival at discharge | From date of inclusion until discharge date from hospitalization of newborn, up to 6 months
  Neonate survival
Survival at 6 months of age | 6 months after birth
  Neonate survival
Oxygen dependence | 6 months after birth

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Gael CORDIER, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris; Nicolas SANANES, MD, PhD, Study Chair — University Hospital, Strasbourg, France; Alexandra BENACHI, MD, PhD, Principal Investigator — AH-HP
Locations (2):
- France (2):
  - Hôpital Béclère, Clamart
  - Hôpital Bicêtre, Le Kremlin-Bicêtre

IPD SHARING:
Plan to Share IPD: No